CLINICAL TRIAL: NCT06083142
Title: Fecal Microbiota Transplant for Autobrewery Syndrome
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Elizabeth L. Hohmann, MD, Physician, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023p000579
Record Dates: First submitted 2023-05-02; First posted 2023-10-13 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-01

CONDITIONS: Auto-Brewery Syndrome; Gut Fermentation Syndrome
Keywords: fecal microbiota transplant
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active FMT (Experimental): Active FMT (5 doses) over 7 days. Each dose contains 15 capsules.
  Interventions: Biological: Fecal microbiota transplantation capsules

INTERVENTIONS:
Biological: Fecal microbiota transplantation capsules — Fecal microbiota transplantation capsules

SUMMARY:
The goal of this clinical trial is to study fecal microbiota transplantation(FMT) by oral capsule in people already diagnosed with auto-brewery syndrome (ABS, also known as gut fermentation syndrome). The main question it aims to answer: Is FMT safe and feasible in this syndrome?

Participants will

1. have a "gut cleanout" with oral antibiotics and a colon cleanse, similar to that administered before colonoscopy
2. receive five oral doses of fecal transplant capsules over a week
3. be followed for six months for safety and research samples

DETAILED DESCRIPTION:
The study is a single arm, open label pilot safety and feasibility study. Subjects will provide medical information related to their diagnosis of ABS. All subjects will have a baseline assessment (medical history, exam, blood and stool samples ) at Massachusetts General Hospital in Boston. Those enrolled will receive a gut clean out procedure and 5 doses of FMT capsules in the 7 days after the clean out. Each individual ABS patient will receive capsules generated from a single donor, to minimize the risk of transmission of infectious agents. All subjects receive active treatment; there is no placebo.

The primary objective of this study is to evaluate the safety and feasibility of the proposed procedures (antibiotic pretreatment, "clean out" and microbial restoration via capsule FMT), thus the primary endpoints will be collection of data regarding any FMT-related adverse events. Feasibility will be defined as taking 3 doses of FMT capsules which we believe can fully reconstitute a healthy microbiome based upon our and others work.

Safety will be assessed daily for 7 days after FMT, and the intermitently over the 6 months after FMT, using standardized patient report scales and interviews as well as by clinical laboratories (at baseline and 2 weeks 2 months, and 6 months). Feasibility is defined as all subjects completing at least 3/5 planned doses of FMT capsules.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 with documented ABS symptoms for at least one year, including supervised ethanol testing or a positive glucose challenge test in a supervised setting.
* Active ABS including at least 3 flares by either serum or breath alcohol levels in the past year (blood or breath samples)
* Subject's microbiome produces alcohol ex vivo in bioreactor (Schnabl laboratory)
* Willing and able to travel to Boston for in person assessment (modest reimbursement available)
* Willing to stop antifungals, and any other complimentary therapies for ABS, if taking
* Medically able to withstand clean out. If participants are over 60, the subject must have previously tolerated a prior colonoscopic "prep" as part of prior routine care.
* Local physician contact available

Exclusion Criteria:

* Unwilling/unable to swallow large capsules (e.g.esophageal stricture or hiatal hernia)
* Delayed gastric emptying syndrome
* Known chronic aspiration, or chronic nausea/vomiting
* Pregnant (pregnancy testing will be performed in women of childbearing potential; women over 52 with no menses for 12 months will not require testing)
* Patients with an acute active illness or acute exacerbation of underlying comorbid condition.
* Patients on unstable, or increasing immunosuppressive agents including high dose corticosteroids(40 mg prednisone daily or more), calcineurin inhibitors, escalating immunosuppression for organ rejection, active chemotherapy with expected neutropenia, current or neutropenia (ANC <1000) within the last year.
* Patients with decompensated cirrhosis, advanced HIV/AIDS, recent bone marrow transplant, or other severe immunodeficiency.
* Severe food allergy or intolerance (donors are omnivores and do not maintain dietary restrictions)
* Cannot document at least 2 COVID vaccinations. Those refusing all COVID vaccination are not eligible for FMT.
* Ulcerative colitis or Crohn's disease (microbiome manipulation may precipitate a flare of these illnesses).
* Active HIV, hepatitis B or C infection (subjects with prior treated hepatitis C must have undetectable viral load; HIV positive subjects must be receiving anti-retroviral therapy with undetectable viral loads x 1 year minimum, Hepatitis B core antibody positive subjects are allowed if negative HepB surface antigen and antibody)
* Taking warfarin (known to be affected by dietary and microbiome changes). NOACs do not exclude.
* On suppressive antibacterial agents, or expected to receive prophylactic antibacterials within the year, for example a patient with a prosthetic heart valve who routinely receives dental prophylaxis, or patient with chronic UTIs anticipated to need treatment frequently
* Known biliary structural abnormalities.
* Allergy to erythromycin, neomycin, or rifaximin.
* Type I diabetes mellitus
* History of pancreatitis or biliary sepsis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Over 6 months.
  Safety outcomes of special interest include:
  Fever, diarrhea, nausea, vomiting, pain/bloating, bacteremia or transmission of GI infection
Adequate dosing of FMT | 7 days
  Adequate dosing is defined as subjects completed the gut cleanse and ingesting at least 3/5 planned doses of FMT capsules

SECONDARY OUTCOMES:
Blood Alcohol Level | Over 6 months
  Plasma blood alcohol level
Stool bioreactor ethanol production | Over 6 monthis
  Presence or absence of elevated alcohol level when stool is cultured in a bioreactor
weight | over 6 months
  Subject weight in kg
Microbiome analysis of stool samples | over 6 months.
  Comparison of stool microbiome to subject's baseline and donor

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hohmann, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
coded data will be shared upon request
Supporting Information: Study Protocol, ICF, CSR
Time Frame: At completion of study
Access Criteria: upon request